CLINICAL TRIAL: NCT05943236
Title: Assessment of the Ankle Joint Axis Using a Long Ankle View Radiograph
Acronym: LAVIEW
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Markus Knupp (Other)
Collaborators: Basel Academy for Quality and Research in Medicine (Unknown); Merian Iselin Klinik (Other)
Responsible Party: Sponsor-Investigator, Markus Knupp, Prof. Dr., Mein Fusszentrum AG
Organization: Mein Fusszentrum AG (Other)
Other Study IDs: LAVIEW
Record Dates: First submitted 2023-05-10; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: X-ray

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients: All patients
  Interventions: Device: Radiographic assessment of the medial-distal tibial angle

INTERVENTIONS:
Device: Radiographic assessment of the medial-distal tibial angle — A long ankle view will be generated within a standard radiographic assessment and the medial-distal tibial angle will be assessed.

SUMMARY:
The study is a reliability (reproducibility) study on a single measurement procedure. Reliability (reproducibility) will be assessed by repeating the whole measurement procedure twice. The measurement procedure studied is the generation of a long ankle view image based on a radiographic assessment followed by a manual assessment of the medial-distal tibial angle.

DETAILED DESCRIPTION:
The study is a reliability (reproducibility) study on a single measurement procedure. Reliability (reproducibility) will be assessed by repeating the whole measurement procedure twice. The measurement procedure studied is the generation of a long ankle view image based on a radiographic assessment followed by a manual assessment of the medial-distal tibial angle (MDTA).

In order to assess the value of different assessment methods of the MDTA, several variants will be considered, which are all applied to the same long ankle view image. To determine the intra- and interrater reliability of the manual assessment, this assessment will be done twice by different observers (one doctoral student, one radiologist) and repeated within each observer.

ELIGIBILITY:
Inclusion

* Clinical indication for a radiographic assessment of the lower half of one leg
* Age above 20

Exclusion Criteria:

* Previous bony procedures (surgery), fractures or anomalies of the lower leg, which does not allow a reliable assessment of the MDTA
* Symptomatic or clinically obvious malalignment at any level of the lower extremity
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical indication for a radiographic assessment of the lower half of one leg
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
medial-distal tibial angle | Day 1 (There is only one single day of contact for each patient)
  The angle is determined based on determining the mechanical axis and the angle axis.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Knupp, MD, Principal Investigator — Praxis "Mein Fusszentrum"
Locations (1):
- Praxis "Meim Fusszentrum", Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data will be provided together with the publication
Supporting Information: Study Protocol
Time Frame: Data will be made available at the date of publication for ever.
Access Criteria: There will be no criteria.